CLINICAL TRIAL: NCT06584526
Title: Effects of Aerobic and Strength Exercice on Nociplastic Pain in Patients with Temporomandibular Disorders: a Randomized Controlled Trial.
Brief Title: Effects of Aerobic and Strength Exercice on Nociplastic Pain in Temporomandibular Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Flora Dantony, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIS-2024-05
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Temporomandibular Disorders (TMD); Nociplastic Pain; Aerobic Exercise; Strengthening Exercises; Myofascial Pain Dysfunction Syndrome, Temporomandibular Joint
MeSH Terms: conditions — Temporomandibular Joint Disorders; Nociplastic Pain; Temporomandibular Joint Dysfunction Syndrome | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physical Therapy (PT) (Active Comparator): 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions (same programme than the experimental groups).
  Education: a series of recommendations to correct inappropriate behaviors such as parafunctions.
  Manual therapy:
  * Bilateral myofascial pressure of 60'' applied to the masseter, temporalis, sternocleidomastoid, and upper trapezius muscles.
  * Dorsal glinding of the Occipital-Atlas segment, performed at Grade III intensity (3sets of 30'', with 15'' of rest).
  Therapeutic exercise:
  * Controlled opening and closing of the jaw: 6 repetitions with 30'' of rest
  * Isometric exercices of the jaw in opening, protrusion, and lateral excursion:3 sets of 10'' for each movement, 15'' of rest
  * Deep neck flexors training using StabilizerTM biofeedback, without contracting the superficial muscles: baseline pressure at 20 mmHg, perform craniocervical flexion at 22, 24, 26, 28, and 30 mmHg, 10'' per stage).
  Interventions: Other: Physical Therapy
- Physical Therapy and Aerobic Exercise (PT+AE) (Experimental): Physical therapy combined with aerobic exercise: 30 minutes of physical therapy (same programme than the other experimental group and the active comparator), combined with a 30 minutes aerobic exercise programme on a cycle ergometer.
  The AE will consist of:
  * Warm-up: Participants cycled for 5 min at a heart rate reserve (HRR) of 50%.
  * Main work: For 24 min, participants performed an interval exercise divided into four intervals, with 4 min at 85%* of the HRR and 2 min of recovery at 50-60% of the HRR in each cycle.
  * Active recovery: The last minute allowed participants to engage in active recovery at 50% of the HRR.
    *: The value of the higher HHR will be reached through a weekly progression:
  * Week 1: 65% HHR
  * Week 2: 70% HHR
  * Week 3: 75% HHR
  * Week 4: 80% HHR
  * Week 5-6: 85% HHR
  The HRR was calculated using the Karvonen formula used in similar studies:
  HRtarget = [HHR x %intensity] + HRrest
  HRR = HRmax - HRrest HRmax = 207 - (0.7 x age)
  HR assessed with a Polar10 sensor.
  Interventions: Other: Physical Therapy and Aerobic Exercise
- Physical Therapy and Strength Exercise (PT+ST) (Experimental): Physical therapy combined with aerobic exercise: 30 minutes of physical therapy (same programme than the other experimental group and the active comparator), combined with a 30 minutes strength exercise (ST) programme.
  The ST exercise will consist of:
  * Warm-up (5'): circuit, 3 sets of: jumping jacks (20''), mountain climbers (20''), abdominal crunch (20''), active stretching of the quadriceps (20'').
  * Main work: For 24 min, a circuit of multiarticular exercise (body weight). Four cycles of 4' of work, with 2' of rest between them. Each exercise will have a work time of 30'' guided with a timer. Intensity will be increased each 2 weeks (W) (higher difficulty and speed).
    * Lunge: W1-2 bilateral 10x / W3-4 unilateral 12x / W5-6 walking 14x
    * Push up: W1-2 inclined 8x / W3-4 normal 10x / W5-6 declined 10x
    * Squat: W1-2 normal 10x / W3-4 lateral lunge 12x / W5-6 step up 10x
    * Core: W1-2 front plank 10x / W3-4 up and down plank 12x / W5-6 superman 12x
  * Active recovery: Walk for 1'.
  Interventions: Other: Physical Therapy and Strength Exercise

INTERVENTIONS:
Other: Physical Therapy — 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions (same programme than the experimental groups).
  Arms: Physical Therapy (PT)
Other: Physical Therapy and Aerobic Exercise — 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions, combined with a 30 minutes aerobic exercise programme on a cycle ergometer.
  Arms: Physical Therapy and Aerobic Exercise (PT+AE)
Other: Physical Therapy and Strength Exercise — 30 minutes of physical therapy with education, manual therapy and therapeutic exercise at both temporomandibular and cervical regions, combined with a 30 minutes strength exercise programme.
  Arms: Physical Therapy and Strength Exercise (PT+ST)

SUMMARY:
Chronic temporomandibular disorders are common in the general population. Nociplastic pain seems to be present in this pathology, with an hypersensitivity to touch, pressure and movement observed in both local and remote areas, as weel as comorbidities such as fatigue, sleep disturbance, difficulty to focus attention and memory disturbance. The best evidence-based treatment of temporomandibular disorders consists in combining education, manual therapy and therapeutic exercise in both temporomandibular and cervical regions. Aerobic and strength exercises showed to be effective in subjects with chronic pain and nociplastic pain, by inducing an hypoalgesic effect. However, there isn't investigation about the effects of theses types of exercise in subjects with temporomandibular disorders and nociplastic pain. Thus, the aim of the study is to determine if adding aerobic or strength exercise to an effective physical therapy programme is more effective than physical therapy alone to improve nociplastic pain in subjects with temporomandibular disorders.

DETAILED DESCRIPTION:
Introduction: Temporomandibular disorders used to improve with education manual therapy and therapeutic exercise. However, despite the evidence oh nociplastic pain in these patients, the treatments remain local. As aerobic and strength exercice have hypoalgesic effect in chronic musculoskeletal pain, we aim to study the effects combined with a common physical therapy programme on nociplastic pain in patients with temporomandibular disorders.

Main objective: Determine if aerobic exercice and strength exercice combined with physical therapy are more effective than physical therapy alone to improve local and remote pressure pain threshold (temporals, masseters, sternocledomastoids, upper trapezius, handgrip, quadriceps and gastrocnemius), in subjects with temporomandibular disorders and nociplastic pain.

Material and methodos:

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a myogenic temporomandibular disorder (DC/TMD) by an odontologist.
* Chronic pain (>3months)
* Nociplastic pain
* Positive Flexion Rotation Test
* Be physically able to realize aerobic and strength exercise (functional movement test)

Exclusion Criteria:

* History of trauma, TMJ or cervical fracture the past three months
* History of TMJ or cervical surgery
* Systemic, rheumatic, metabolic, neurologic, psychiatric, pulmonary diseases or neoplastic malignant
* History of cardiovascular diseases which contraindicate aerobic exercise
* Current orthodontic treatment, splints for bruxism
* Drug addiction, alcoholism
* Pregnancy
* Use of analgesic medication less than 48 hours before each data collection
* Physical therapy treatment during the past three month

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-09-09 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of baseline in Pain Pressure Threshold at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Bilateral measure with digital algometer, applying a perpendicular pressure of 0.5 kg/cm2/s on: masseter, temporal, upper trapezius, SCOM, quadriceps tendon, achilles Tendon.

SECONDARY OUTCOMES:
Change of baseline in Jaw function at 6 weeks (final) and 12 weeks (post) | Baseline - 1 month (final) - 3 months
  Fonseca Anamnestic Index. 10 questions with a three-point scale: 0 = no, 5 = sometimes and 10 = yes; total score from 0 good function, to 100 worst.
Change of baseline in Strength at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Handgrip strength will be assessed with a Jamar dynamometer, maximal isometric strength, 2 times.
  Maximal strength of upper trapezius, quadriceps and gastrocnemius will be assessed with a digital dynamometer ActivForce, maximal isometric strength, 2 times.
  Before assessing strength, a 10 minutes warm up of the muscles will be done:
  * Upper trapezius: shoulder elevations
  * Quadriceps: squat
  * Gastrocnemius: heel elevations
  * Handgrip: press a ball
Change of baseline in Upper Cervical ROM at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Assessment of upper cervical ROM performing the Flexion Rotation Test with a CROM device.
Change of baseline in Central Sensitization at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Central Sensitization Index: 25 items, from 0 to 100 (0-29=subclinic; 30-39=mild; 40-59=moderate; 60-100=extrem)
Change of baseline in Rest Heart Rate at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Patient sitting for 5 minutes to rest, and then heart rate is assessed with a Polar H10 sensor.
Change of baseline in Anxiety and depression at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Hospital Anxiety and Depression Scale: 2 subscales, one for anxiety and the other one for depression. Each scale score is from 0 (less) to 21 (worst)
Change of baseline in Sleep Quality at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Pittsburgh Sleep Quality Index: maximum score of 21; 5 being the cut-off point.
Change of baseline in Kinesiophobia at 6 weeks (final) and 12 weeks (post) | Baseline - 6 weeks (final) - 12 weeks
  Tampa Scale of Kinesiophobia: from 10 to 40 (Likert scale 4 points: 1 = totally disagree; 2 = disagree; 3 = agree; 4 = totally agree). Cut-off: 23.
Adherence at 6 weeks (final) and 12 weeks (post) | 6 weeks (final) - 12 weeks
  ATTEMPT questionnaire to evaluate adherence to exercises post-intervention. 6 items, Likert scale 5 punts ( 1 = totally disagree; 2 = disagree; 3 = neutral; 4 = agree; 5 = totally agree). From 6 to 30, a change of 4 indicates a change.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided